CLINICAL TRIAL: NCT06515470
Title: A First-in-Human, Open-Label, Dose Escalation and Expansion Trial of BTX-9341 in Participants With Advanced and/or Metastatic Breast Cancer
Brief Title: Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BTX-9341 in Advanced and/or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biotheryx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTX-9341-101
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: HR+/HER2-
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- BTX-9341 (Part A) (Experimental): BTX-9341 capsule(s) administered orally once daily (QD) in 28-day cycles
  Interventions: Drug: BTX-9341
- BTX-9341 + fulvestrant (Part A) (Experimental): BTX-9341 capsule(s) administered orally QD in 28-day cycles and fulvestrant intermuscular injections on Day 15 and then once every 28 days
  Interventions: Drug: BTX-9341; Drug: Fulvestrant
- BTX-9341 + fulvestrant (Part B) (Experimental): BTX-9341 capsule(s) administered orally QD in 28-day cycles and fulvestrant intermuscular injections on Day 15 and then once every 28 days
  Interventions: Drug: Fulvestrant; Drug: BTX-9341

INTERVENTIONS:
Drug: BTX-9341 — Daily oral dose in 28-day cycles until maximum tolerated dose (MTD) or maximum evaluable dose (MED) determined
  Arms: BTX-9341 (Part A); BTX-9341 + fulvestrant (Part A)
Drug: Fulvestrant — 500 mg intramuscular injections on Day 15 and then every 28 days
  Other Names: Faslodex
  Arms: BTX-9341 + fulvestrant (Part A); BTX-9341 + fulvestrant (Part B)
Drug: BTX-9341 — Daily oral dose in 28-day cycles using dose determined in Part A
  Arms: BTX-9341 + fulvestrant (Part B)

SUMMARY:
The purpose of this study is to test BTX-9341 alone or in combination with fulvestrant (a currently marketed medication for breast cancer) in participants with advanced and/or metastatic hormone receptor positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) breast cancer. The study includes a dose escalation part (Part A) where small groups of participants will receive increasing doses of BTX-9341 or BTX-9341 + fulvestrant followed by a dose expansion part (Part B) where participants will receive the dose of BTX-9341 selected in Part A + fulvestrant.

DETAILED DESCRIPTION:
This first-in-human (FIH), Phase 1 study of BTX-9341 is multicenter, nonrandomized, and open-label to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of BTX-9341 in participants with advanced and/or metastatic HR+/HER2 breast cancer. The study will include a dose escalation part (Part A) followed by a dose expansion part (Part B). During Part A, BTX-9341 will initially be dose escalated alone and then in combination with fulvestrant. A single combination therapy cohort of BTX-9341 + fulvestrant will be further explored in Part B. BTX-9341 will be administered orally in 28-day treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic and/or locally advanced HR+/HER2- breast cancer (dose escalation: measurable disease and/or at least 1 lytic or mixed [lytic + sclerotic] bone lesion that can be assessed by CT or MRI or non-measurable disease [including bone lesions]; dose expansion: measurable disease)
* Dose escalation: (a) received not more than 1 chemotherapy in the metastatic/advanced setting; (b) no limit to the lines of endocrine therapy (monotherapy or combination therapy) in the metastatic setting; (c) received CDK4/6 inhibitor therapy
* Dose expansion: (a) received not more than 1 chemotherapy in metastatic/advanced setting; (b) received not more than 2 lines of endocrine therapy (monotherapy or combination therapy) and must have been on prior endocrine therapy for at least 6 months before progression; (c) received at most 2 lines of CDK4/6 inhibitor therapy (1 in the adjuvant setting and 1 in the metastatic setting) and must have been on prior CDK4/6 inhibitor therapy for at least 6 months
* Acceptable hematologic function

  1. ANC ≥ 1500 per mL. Note: Use of growth-factors to maintain the ANC criterion is prohibited.
  2. Platelet count ≥ 100,000 per mL. Note: Use of transfusions or thrombopoietic agents to achieve the baseline platelet count criterion is prohibited.
  3. Hemoglobin ≥ 9.0 g/dL. Note: Packed red blood cell transfusion is allowed up to 14 days prior to trial entry.
* Acceptable liver function

  1. Bilirubin ≤ 2.0 × institutional upper limit of normal (ULN) (or < 3.0 × institutional ULN if Gilbert's disease is present)
  2. Alanine transaminase (ALT)/aspartate aminotransferase (AST) ≤ 3.0 × institutional ULN (≤ 5.0 × institutional ULN if liver metastases present)
  3. Alkaline phosphatase ≤ 2.5 × institutional ULN (≤ 5.0 × institutional ULN if bone or liver metastases present)
* Able and willing to sign informed consent
* Meets all study requirements in the opinion of the Investigator

Exclusion Criteria:

* RB1 (retinoblastoma) gene mutation
* Symptomatic visceral disease
* Clinical evidence or history of central nervous system metastasis
* Abnormalities in coagulation, such as bleeding diathesis, or treatment with anticoagulants precluding injections of fulvestrant or luteinizing hormone-releasing hormone (LHRH) agonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of BTX-9341 | Up to 28 days after last dose of BTX-9341
  Frequency and severity, incidence of treatment-emergent and treatment-related adverse events using NCI-CTCAE v5.0
Part A: Number of Participants With Dose Limiting Toxicities (DLTs) | 28 days
  DLT rate in Cycle 1
Part A: Determine MTD/MED of BTX-9341 in monotherapy | Approximately 1 year from study start
  Based on CTCAE v5.0 assessment of adverse events
Part A: Determine MTD/MED of BTX-9341 in combination therapy | Approximately 18 months from study start
  Based on CTCAE v5.0 assessment of adverse events
Part B Combination Therapy: Objective Response (OR) rate | Approximately 18 months from start of Part B
  OR is the confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 as determined by Investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Barton, MD, Study Director — Chief Medical Officer
Locations (6):
- United States (6):
  - Biotheryx Investigative Site, Rochester, Minnesota
  - Biotheryx Investigative Site, Omaha, Nebraska
  - Biotheryx Investigative Site, Houston, Texas
  - Biotheryx Investigative Site, San Antonio, Texas
  - Biotheryx Investigative Site, West Valley City, Utah
  - Biotheryx Investigative Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No